CLINICAL TRIAL: NCT01237080
Title: Intubation of Morbidly Obese Patients. A Randomized Clinical Trial, Comparing GlideScope ® With Fastrach TM.
Brief Title: Intubation of Morbidly Obese Patients. A Clinical Trial, Comparing Glide Scope ® With Fastrach TM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Mogens Ydemann Nielsen, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-1-2010-058
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-01

CONDITIONS: Morbidly Obese; Intubationtime; Intubationattempts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fastrach (Experimental): 50 persons beeing intubated using the Fastrach.
  Interventions: Device: Fastrach
- GlideScope (Experimental): 50 persons beeing intubated using the GlideScope.
  Interventions: Device: GlideScope

INTERVENTIONS:
Device: GlideScope — The GlideScope is an anatomically shaped, rigid, fibreoptic videolaryngoscope.
  Arms: GlideScope
Device: Fastrach — The Fastrach is an intubation laryngeal mask.
  Arms: Fastrach

SUMMARY:
The purpose of this study is to compare the GlideScope ® and the Fastrach TM for intubation of morbidly obese. Mainly we will try to clarify which of the instruments that produce the shortest intubationtime and lowest number of intubationattempts.

The hypothesis is that intubation would be 1) quicker and 2) with the lowest number of attempts, using the GlideScope®.

DETAILED DESCRIPTION:
The number of obese people rises. Thus 25.2% of Danish 9th graders are obese. As a result, surgery and anesthesia in obese patients becomes more frequent. Several potential problems related to anesthesia in this patient group exists, including airway management and sufficient oxygenation.

Anaesthesia of obese patients are more likely to require intubation. In light of the foregoing, it is therefore important to find the methods that provide the fewest complications related to intubation. Therefore this study compare two instruments (Fastrach TM and GlideScope ®) to find out which of the methods that provides the best airway management, measured primarily in time and numbers of intubation attempts.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/= 35

Exclusion Criteria:

* need for crash induction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogens VY Nielsen, MD, Principal Investigator — Department of Anesthesiology, Copenhagen University Hospital, Glostrup, Denmark
Locations (2):
- Denmark (2):
  - Department of Anesthesiology, Copenhagen University Hospital, Glostrup Municipality, Zeeland
  - Privathospitalet Hamlet, Soeborg, Zeeland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from September 2010 to January 2011. Patients were recuted from two hospitals.
Pre-assignment Details: Exclusion: severe mental disorder, greater alcohol consumption than recommended by the Danish Health Authority, drug abuse, previously impossible mask ventilation or intubation with the GS and/or FT, the need for RSI and if the anaesthetist responsible determined that the patient should be treated differently than described in the protocol.
Period: Overall Study
Arm/Group | Fastrach | GlideScope
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fastrach | GlideScope | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Full Range); unit: years] | 42 (NA) [19 to 59] | 43 (NA) [19 to 60] | 42 (999999) [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 43 | 76
  Male | 17 | 7 | 24
Region of Enrollment [Number; unit: participants]
  Denmark | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Intubated in the First Attempt
Description: The intubation attempt was considered a failure if the GS or the FT was removed from the patient's mouth and required reinsertion or if the cuff had been inflated and the tube needed to be replaced (e.g., in oesophageal intubation).
Time Frame: please see description
Measure: Number; unit: participants
Arm/Group | Fastrach | GlideScope
Number analyzed (Participants) | 50 | 50
participants | 42 | 46

2. Secondary Outcome: Lowest Saturation During Intubation.
Time Frame: measured on the monitor
Reporting Status: Not Posted

3. Secondary Outcome: Mucosal Lesion
Time Frame: inspection during intubation and one hour postop.
Reporting Status: Not Posted

4. Secondary Outcome: Subjectively Intubation Difficulty
Time Frame: measured immediately on a visual analogue scale.
Reporting Status: Not Posted

5. Secondary Outcome: Intubation of the Esophagus.
Time Frame: detected immediately
Reporting Status: Not Posted

6. Secondary Outcome: Postoperative Hoarseness.
Time Frame: one hour postoperative.
Reporting Status: Not Posted

7. Secondary Outcome: Postoperative Throat Pain.
Time Frame: one hour postoperative
Reporting Status: Not Posted

8. Primary Outcome: Time to Intubate
Time Frame: From when the anaesthetist picked up the GS / FT until a typical capnogram was seen on the capnograph.
Population: The sample size was calculated to 40 in each group (50 patients were included in each group): minimum relevant difference in intubation time of 20 s and a standard deviation of 28 s. A significance level of 0.05 and an acceptable risk of Type 2 error of 0.1 were used.
Measure: Mean (95% Confidence Interval); unit: sec
Arm/Group | Fastrach | GlideScope
Number analyzed (Participants) | 50 | 50
sec | 61 [46 to 76] | 49 [40 to 57]

ADVERSE EVENTS:
Arm/Group | Fastrach | GlideScope
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Acta Anaesthesiol Scand 2012; 56: 755-761

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No